CLINICAL TRIAL: NCT04292730
Title: A Phase 3 Randomized Study to Evaluate the Safety and Antiviral Activity of Remdesivir (GS-5734™) in Participants With Moderate COVID-19 Compared to Standard of Care Treatment
Brief Title: Study to Evaluate the Safety and Antiviral Activity of Remdesivir (GS-5734™) in Participants With Moderate Coronavirus Disease (COVID-19) Compared to Standard of Care Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-540-5774; 2020-000842-32 (EudraCT Number); ISRCTN85762140 (Other: ISRCTN)
Expanded Access: NCT04323761 (Approved for marketing)
Record Dates: First submitted 2020-02-28; First posted 2020-03-03 (Actual); Results first posted 2021-01-26 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — remdesivir; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part A: Remdesivir (RDV), 5 Days (Experimental): Participants will receive continued standard of care (SOC) therapy together with RDV 200 mg on Day 1 followed by RDV 100 mg on Days 2, 3, 4, and 5.
  Interventions: Drug: Remdesivir; Drug: Standard of Care
- Part A: Remdesivir, 10 Days (Experimental): Participants will receive continued standard of care therapy together with RDV 200 mg on Day 1 followed by RDV 100 mg on Days 2, 3, 4, 5, 6, 7, 8, 9, and 10.
  Interventions: Drug: Remdesivir; Drug: Standard of Care
- Part A: SOC Therapy (Active Comparator): Participants will receive continued standard of care therapy.
  Interventions: Drug: Standard of Care
- Part B: Extension Treatment, Remdesivir 10 Days (Experimental): Participants will receive continued standard of care therapy together with RDV 200 mg on Day 1 followed by RDV 100 mg on Days 2, 3, 4, 5, 6, 7, 8, 9, and 10.
  Interventions: Drug: Remdesivir; Drug: Standard of Care

INTERVENTIONS:
Drug: Remdesivir — Administered as an intravenous infusion
  Other Names: GS-5734™; Veklury®
  Arms: Part A: Remdesivir (RDV), 5 Days; Part A: Remdesivir, 10 Days; Part B: Extension Treatment, Remdesivir 10 Days
Drug: Standard of Care — Standard of Care Treatment for COVID-19 Infection

SUMMARY:
The primary objective of this study was to evaluate the efficacy of 2 remdesivir (RDV) regimens compared to standard of care (SOC), with respect to clinical status assessed by a 7-point ordinal scale on Day 11.

ELIGIBILITY:
Key Inclusion Criteria:

* Willing and able to provide written informed consent prior to performing study procedures (participants ≥ 18 years of age) or assent (participants ≥ 12 and < 18 years of age) prior to performing study procedures. For participants ≥ 12 and < 18 years of age, a parent or legal guardian willing and able to provide written informed consent prior to performing study procedures
* Severe Acute Respiratory Syndrome Coronavirus (SARS-CoV)-2 infection confirmed by polymerase chain reaction (PCR) test ≤ 4 days before randomization
* Currently hospitalized and requiring medical care for COVID-19
* Peripheral capillary oxygen saturation (SpO2) > 94% on room air at screening
* Radiographic evidence of pulmonary infiltrates

Key Exclusion Criteria:

* Participation in any other clinical trial of an experimental treatment for COVID-19
* Concurrent treatment or planned concurrent treatment with other agents with actual or possible direct acting antiviral activity against SARS-CoV-2
* Requiring mechanical ventilation at screening
* Alanine Aminotransferase (ALT) or aspartate aminotransferase (AST) > 5 X upper limit of normal (ULN)
* Creatinine clearance < 50 mL/min using the Cockcroft-Gault formula for participants ≥ 18 years of age {Cockcroft 1976} and Schwartz Formula for participants < 18 years of age

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1113 (Actual)
Dates: Start 2020-03-15 (Actual); Primary Completion 2020-04-29 (Actual); Study Completion 2020-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (183):
- United States (106):
  - Kaiser Permanente Los Angeles Medical Center, 3340 E. La Palma Avenue, Anaheim, California
  - Alta Bates Summit Medical Center, Berkeley, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - Eden Medical Center, Castro Valley, California
  - Kaiser Permanente Los Angeles Medical Center, 9333 Imperial Highway, Downey, California
  - Kaiser Permanente Los Angeles Medical Center, 9961 Sierra Ave, Fontana, California
  - St Joseph Hospital Eureka, Fortuna, California
  - Kaiser Permanente Los Angeles Medical Center, 25825 S. Vermont Ave., Harbor City, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Kaiser Permanente Los Angeles Medical Center, 6041 Cadillac Ave., Los Angeles, California
  - Kaiser Permanente Los Angeles Medical Center, 5601 De Soto Avenue, Los Angeles, California
  - Mission Hospital Regional Medical Center, Mission Viejo, California
  - Kaiser Permanente Los Angeles Medical Center,27300 Iris Avenue, Moreno Valley, California
  - El Camino Hospital, Mountain View, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Kaiser Permanente Oakland Medical Center, Oakland, California
  - Kaiser Permanente Los Angeles Medical Center, 2295 S. Vineyard Avenue, Ontario, California
  - The Center for Cancer Prevention and Treatment at St. Joseph Hospital of Orange, Orange, California
  - Kaiser Permanente Los Angeles Medical Center,13651 Willard Street, Panorama City, California
  - Kaiser Permanente Los Angeles Medical Center, 10800 Magnolia Avenue, Riverside, California
  - Sutter Medical Center Sacramento, One Medical Plaza, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - Kaiser Permanente Los Angeles Medical Center, 4647 Zion Avenue, San Diego, California
  - Kaiser Permanente Los Angeles Medical Center, 9455 Clairemont Mesa Blvd, San Diego, California
  - Kaiser Permanente Oakland Medical Center, 1200 El Camino Real, San Francisco, California
  - California Pacific Medical Center-Infectious Disease Associates Medical Group, San Francisco, California
  - Kaiser Permanente Oakland Medical Center, 2425 Geary Blvd, San Francisco, California
  - Kaiser Permanente Oakland Medical Center, 250 Hospital Parkway, Suite 850, San Jose, California
  - Kaiser Permanente Oakland Medical Center, 2500 Merced St, San Leandro, California
  - Kaiser Permanente Oakland Medical Center, 700 Lawrence Expressway, Santa Clara, California
  - Providence St. Johns Medical Center, Santa Monica, California
  - Sutter Santa Rosa Regional Hospital, Santa Rosa, California
  - Stanford Hospital, Stanford, California
  - University of Colorado Denver, University of Colorado Hospital, Aurora, Colorado
  - SCL Health St. Joseph Hospital, 1375 East 19th Ave, Denver, Colorado
  - SCL Health St. Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - SCL Health St. Joseph Hospital, 200 Exempla Circle., Lafayette, Colorado
  - Yale University, New Haven, Connecticut
  - Kaiser Permanente Hawaii Moanalua Medical Center, Honolulu, Hawaii
  - Cook County General Hospital, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - IU Health Methodist Hospital, Indianapolis, Indiana
  - University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - Tulane University, New Orleans, Louisiana
  - Maine Medical Center, Portland, Maine
  - Holy Cross Hospital, Silver Spring, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Brigham & Women's Hospital and Harvard Medical School, Boston, Massachusetts
  - Center for Virology and Vaccine Research, Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - The University of Michigan Hospitals and Health Systems, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Hennepin Healthcare, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Providence St Patrick Hospital and International Heart Institute of MT Foundation, Missoula, Montana
  - Darmouth-Hitchhock Medical Center, Lebanon, New Hampshire
  - Hackensack Medical Center, Hackensack, New Jersey
  - Robert Wood Johnson University Hospital Somerset, Hillsborough, New Jersey
  - Robert Wood Johnson University Hospital Somerset, 1 RWJ Place, New Brunswick, New Jersey
  - Robert Wood Johnson University Hospital Somerset, 201 Lyons Avenue, Newark, New Jersey
  - St. Joseph's University Medical Center, Paterson, New Jersey
  - Jamaica Hospital Medical Center, Jamaica, New York
  - Danbury Hospital, Lagrangeville, New York
  - North Shore University Hospital, Manhasset, New York
  - North Shore University Hospital, 270-05 76th Ave, New Hyde Park, New York
  - Icahn School of Medicine at Mount Sinai, 350 East 17th Street, New York, New York
  - Icahn School of Medicine at Mount Sinai, 1000 10th Avenue, New York, New York
  - Icahn School of Medicine at Mount Sinai, 440 West 114th St., New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Columbia University Irving Medical Center, New York, New York
  - Weill Cornell Medical College/NYU Presbyterian Hospital, New York, New York
  - Jacobi Medical Center, The Bronx, New York
  - James J. Peters Veterans Administration Medical Center, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Kaiser Sunnyside Medical Center, 2875 NW Stucki Ave, Hillsboro, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Kaiser Sunnyside Medical Center, Portland, Oregon
  - Hospital of the University of Pennsylvania, 51 N. 31st Street, Philadelphia, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - The Miriam Hospital, Providence, Rhode Island
  - Prisma Health Richland Hospital, Columbia, South Carolina
  - Prisma Health Richland Hospital, 701 Grove Road, Greenville, South Carolina
  - The Liver Institute of Methodist Dallas Medical Center, Dallas, Texas
  - UT Southwestern Medical Center Amelia Court, HIV Research Clinic, Dallas, Texas
  - Baylor University Medical Center, Dallas, Texas
  - UT Southwestern Medical Center Amelia Court, HIV Research Clinic, 5201 Harry Hines Blvd., Dallas, Texas
  - UT Southwestern Medical Center Amelia Court, HIV Research Clinic, 6201 Harry Hines Blvd, Dallas, Texas
  - Baylor University Medical Center, 1400 8th Ave, Fort Worth, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Baylor University Medical Center, 2401 S. 31st St., Temple, Texas
  - University of Utah Health, Salt Lake City, Utah
  - Virginia Hospital Center, Arlington, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - VCU Health Medical Center, Richmond, Virginia
  - Providence Medical Research Center, Everett, Washington
  - Kadlec Regional Medical Center, Kennewick, Washington
  - Providence St. Peter Hospital, Olympia, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Swedish Center for Comprehensive Care, Seattle, Washington
  - MultiCare Deaconess Hospital, Spokane, Washington
  - MultiCare Tacoma General Hospital, Tacoma, Washington
  - St Joseph Medical Center, Tacoma, Washington
- The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, China
- France (5):
  - CHU Pellegrin, Bordeaux
  - CHU de Montpellier-Hopital Gui de Chauliac, Montpelier Cedex 5
  - CHU de Nantes-Hotel Dieu, Nantes
  - Hopital Saint-Louis, Paris
  - Hopital Saint Antoine, Paris
- Germany (8):
  - Charite Universitatsmedizin Berlin, Campus Virchow-Klinikum, Medizinische Klinik Infektiologie Pneumologie, Berlin
  - Universitatsklinikum Dusseldorf, Klinik fur Gastroenterologie, Hepatologie und Infektiologie, Düsseldorf
  - Universitatsklinikum Hamburg-Eppendorf, Hamburg
  - Universitätsklinikum Schleswig-Holstein Campus Kiel, Kiel
  - Klinikum St. Georg gGmbH Klinik fur Infektiologie, Tropenmedizin, Nephrologie und Rheumatologie, Leipzig
  - Klinikum rechts der Isar der TU Munchen, Klinik und Poliklinik Innere Medizin 2, Munich
  - Klinik für Hämatologie, Onkologie, Immunologie, München
  - Robert-Bosch-Krankenhaus (RBK), Klinik Schillerhohe (KSH) und Dr. Margarete Fischer-Bosch-Institut fur klinische Pharmakologie (IKP), Stuttgart
- Hong Kong (3):
  - Prince of Wales Hospital, Hong Kong
  - Princess Margaret Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong
- Italy (12):
  - UOC Malattie Infettive, ASST Papa Giovanni XXIII, Bergamo
  - ASST degli Spedali Civili di Brescia, Brescia
  - ASST di Cremona - Azienda Socio Sanitaria Territor, Cremona
  - UO Malattie Infettive, Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - UOC Malattie Infettive, IRCCS Ospedale San Raffaele, Milan
  - ASST Fatebenefratelli Sacco, Milan
  - UOC Malattie Infettive e Tropicali, Azienda Ospedaliera di Padova, Padova PD
  - Azienda Ospedaliero Universitaria di Parma, Parma
  - Malattie Infettive I, Fondazione IRCCS Policlinico San Matteo, Pavia
  - Ospedale Guglielmo da Saliceto AUSL di Piacenza, Piacenza
  - UOC Malattie Infettive ad Alta Intensita di Cure, Istituto Nazionale Malattie Infettive Lazzaro Spallanzani I.R.C.C.S., Roma
  - Clinica Universitaria Malattie Infettive, Ospedale Amedeo di Savoia, Torino
- Japan (3):
  - Yokohama Municipal Citizen's Hospital, Kanagawa
  - Nagoya City East Medical Center, Nagoya
  - Tokyo Metropolitan Bokutoh Hospital, Tokyo
- Netherlands (3):
  - Amsterdam University Medical Centre - Location AMC, Amsterdam
  - Leiden University Medical Center, Leiden
  - Erasmus Medical Centre, Rotterdam
- Singapore (3):
  - National University Hospital, Singapore
  - Singapore General Hospital, Singapore
  - National Centre for Infectious Diseases, Tan Tock Seng Hospital, Singapore
- South Korea (3):
  - Kyungpook National University Hospital, Daegu
  - Seoul Medical Center, Seoul
  - National Medical Center, Seoul
- Spain (13):
  - Hospital Principe de Asturias, Alcalá de Henares, Madrid
  - Complejo Hospitalario Universitario A Coruña, A Coruña
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitari de Bellvitge, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario Cruces, Bizkaia
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Regional Universitario de Málaga, Málaga
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitari i Politecnic La Fe, Valencia
- Sweden (3):
  - Sahlgrenska University Hospital, Ostra, Gothenburg
  - SUS (Skanes University Hospital), Malmo
  - Karolinska University Hospital, Stockholm
- Switzerland (3):
  - Hopitaux Universitaires de Genève, Geneva
  - Ospedale Regionale di Locarno La Carità, Lugano
  - Universitätsspital Zürich, Zurich
- Taiwan (3):
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei
- United Kingdom (14):
  - Imperial College NHS Trust, London, Greater London
  - NHS Lothian, Royal lnfirmary of Edinburgh, Edinburgh
  - Queen Elizabeth University Hospital, Glasgow
  - Hull University Teaching Hospitals NHS Trust, Hull
  - Royal Lancaster Hospital, Lancaster
  - Liverpool University Hospital, Liverpool
  - Northwick Park Hospital, London
  - Royal Free London NHS Foundation Trust, London
  - King's College Hospital NHS Trust, London
  - University College London, London
  - Manchester University NHS Foundation Trust, Manchester
  - Pennine Acute Hospitals NHS Trust, Manchester
  - Derriford Hospital, Plymouth
  - Sheffield Teaching Hospitals, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at https://www.gilead.com/science-and-medicine/research/clinical-trials-transparency-and-data-sharing-policy.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: https://www.gilead.com/science-and-medicine/research/clinical-trials-transparency-and-data-sharing-policy

REFERENCES:
- [Result] Spinner CD, Gottlieb RL, Criner GJ, Arribas Lopez JR, Cattelan AM, Soriano Viladomiu A, Ogbuagu O, Malhotra P, Mullane KM, Castagna A, Chai LYA, Roestenberg M, Tsang OTY, Bernasconi E, Le Turnier P, Chang SC, SenGupta D, Hyland RH, Osinusi AO, Cao H, Blair C, Wang H, Gaggar A, Brainard DM, McPhail MJ, Bhagani S, Ahn MY, Sanyal AJ, Huhn G, Marty FM; GS-US-540-5774 Investigators. Effect of Remdesivir vs Standard Care on Clinical Status at 11 Days in Patients With Moderate COVID-19: A Randomized Clinical Trial. JAMA. 2020 Sep 15;324(11):1048-1057. doi: 10.1001/jama.2020.16349. PMID 32821939
- [Derived] Grundeis F, Ansems K, Dahms K, Thieme V, Metzendorf MI, Skoetz N, Benstoem C, Mikolajewska A, Griesel M, Fichtner F, Stegemann M. Remdesivir for the treatment of COVID-19. Cochrane Database Syst Rev. 2023 Jan 25;1(1):CD014962. doi: 10.1002/14651858.CD014962.pub2. PMID 36695483
- [Derived] Ansems K, Grundeis F, Dahms K, Mikolajewska A, Thieme V, Piechotta V, Metzendorf MI, Stegemann M, Benstoem C, Fichtner F. Remdesivir for the treatment of COVID-19. Cochrane Database Syst Rev. 2021 Aug 5;8(8):CD014962. doi: 10.1002/14651858.CD014962. PMID 34350582

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States, Europe, and Asia. The first participant was screened on 15 March 2020. The last study visit occurred on 26 June 2020.
Pre-assignment Details: 1138 participants were screened.
Groups:
- Part A: Remdesivir (RDV) for 5 Days: Participants received continued standard of care (SOC) therapy together with intravenous (IV) RDV 200 mg on Day 1 followed by IV RDV 100 mg on Days 2-5.
- Part A: Remdesivir for 10 Days; Part B: Extension Treatment, Remdesivir for 10 Days: Participants received continued SOC therapy together with IV RDV 200 mg on Day 1 followed by IV RDV 100 mg on Days 2-10.
- Part A: SOC Therapy: Participants received continued SOC therapy.
Period: Overall Study
Arm/Group | Part A: Remdesivir (RDV) for 5 Days | Part A: Remdesivir for 10 Days | Part A: SOC Therapy | Part B: Extension Treatment, Remdesivir for 10 Days
Started | 199 | 197 | 200 | 517
Completed | 179 | 176 | 178 | 437
Not Completed | 20 | 21 | 22 | 80
Not completed — Lost to Follow-up | 8 | 12 | 12 | 48
Not completed — Death | 2 | 2 | 4 | 12
Not completed — Withdrew Consent | 2 | 2 | 5 | 6
Not completed — Non-Compliance with Study Drug | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 0
Not completed — Randomized but not Treated | 8 | 4 | 0 | 14

BASELINE CHARACTERISTICS:
Population: Part A: Safety Analysis Set included participants who were randomized into part A of the study and received at least 1 dose of study treatment or completed the Day 1 visit (SOC only group).
  Part B: Expanded RDV-Treated Analysis Set included participants who were enrolled into Part B of the study and received at least 1 dose of study drug.
Groups:
- Part A: Remdesivir for 5 Days: Participants received continued SOC therapy together with IV RDV 200 mg on Day 1 followed by IV RDV 100 mg on Days 2-5.
- Total: Total of all reporting groups
Arm/Group | Part A: Remdesivir for 5 Days | Part A: Remdesivir for 10 Days | Part A: SOC Therapy | Part B: Extension Treatment, Remdesivir for 10 Days | Total
Number analyzed (Participants) | 191 | 193 | 200 | 503 | 1087
Age, Customized [Count of Participants; unit: Participants]
  Age, Categorical: < 65 Years | 142 | 141 | 142 | 351 | 776
  Age, Categorical: >= 65 Years | 49 | 52 | 58 | 152 | 311
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 75 | 75 | 221 | 448
  Male | 114 | 118 | 125 | 282 | 639
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Not Permitted means local regulators did not allow collection of race information.
  Participants
    Race: American Indian or Alaska Native | 2 | 0 | 1 | 3 | 6
    Race: Asian | 34 | 31 | 37 | 61 | 163
    Race: Black | 35 | 37 | 27 | 107 | 206
    Race: Native Hawaiian or Pacific Islander | 1 | 1 | 1 | 1 | 4
    Race: White | 109 | 107 | 112 | 260 | 588
    Race: Not Permitted | 5 | 5 | 7 | 21 | 38
    Race: Other | 5 | 12 | 15 | 50 | 82
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Not Permitted means local regulators did not allow collection of ethnicity information.
  Participants
    Ethnicity: Hispanic or Latino | 25 | 42 | 34 | 156 | 257
    Ethnicity: Not Hispanic or Latino | 162 | 144 | 152 | 325 | 783
    Ethnicity: Not Permitted | 4 | 7 | 13 | 22 | 46
    Ethnicity: Missing | 0 | 0 | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 76 | 99 | 85 | 318 | 578
  Spain | 37 | 28 | 31 | 44 | 140
  Italy | 30 | 23 | 26 | 54 | 133
  United Kingdom | 7 | 9 | 17 | 27 | 60
  South Korea | 7 | 4 | 10 | 16 | 37
  Germany | 8 | 6 | 8 | 13 | 35
  Singapore | 3 | 6 | 9 | 14 | 32
  Hong Kong | 9 | 11 | 7 | 1 | 28
  Switzerland | 4 | 5 | 6 | 3 | 18
  France | 2 | 1 | 0 | 5 | 8
  Taiwan | 5 | 1 | 0 | 0 | 6
  Netherlands | 3 | 0 | 1 | 1 | 5
  Japan | 0 | 0 | 0 | 4 | 4
  Sweden | 0 | 0 | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Part A: Percentage of Participants in Each Clinical Status Category as Assessed by a 7-Point Ordinal Scale on Day 11
Description: Clinical status was derived from death, hospital discharge, and ordinal scale as follows: score of "1" was used for all days on or after the date of death; score of "7" was used for all days on or after discharged alive date; last available assessment for missing value. The scale is as follows: 1. Death; 2. Hospitalized, on invasive mechanical ventilation or Extracorporeal Membrane Oxygenation (ECMO); 3. Hospitalized, on non-invasive ventilation or high flow oxygen devices; 4. Hospitalized, requiring low flow supplemental oxygen; 5. Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (coronavirus (COVID-19) related or otherwise); 6. Hospitalized, not requiring supplemental oxygen - no longer required ongoing medical care (other than per protocol remdesivir administration; 7. Not hospitalized. The odds ratio represents the odds of improvement in the ordinal scale for a RDV group relative to the SOC group.
Time Frame: Day 11
Population: Full Analysis Set (FAS) included all participants who were randomized into Part A of the study and received at least 1 dose of study treatment if randomized to 1 of the RDV treatment groups. Participants in the SOC arm who had protocol Day 1 visit were included in the FAS.
Measure: Number; unit: percentage of participants
Arm/Group | Part A: Remdesivir for 5 Days | Part A: Remdesivir for 10 Days | Part A: SOC Therapy
Number analyzed (Participants) | 191 | 193 | 200
percentage of participants
  Score: 1 | 0.0 | 1.0 | 2.0
  Score: 2 | 0.0 | 0.5 | 2.0
  Score: 3 | 2.6 | 0.0 | 3.5
  Score: 4 | 3.7 | 6.2 | 5.5
  Score: 5 | 19.9 | 22.8 | 23.0
  Score: 6 | 3.7 | 4.7 | 4.0
  Score: 7 | 70.2 | 64.8 | 60.0
Statistical Analysis 1: Comparison: Part A: Remdesivir for 5 Days vs Part A: SOC Therapy; Primary analysis; Test type: Superiority; p = 0.0174, Proportional odds model — P-value was calculated using proportional odds model with treatment as the independent variable; Odds Ratio (OR) = 1.65, 95% CI 2-sided [1.092 to 2.483]
Statistical Analysis 2: Comparison: Part A: Remdesivir for 10 Days vs Part A: SOC Therapy; Primary analysis; Test type: Superiority; p = 0.1826, Proportional odds model — P-value was calculated using proportional odds model with treatment as the independent variable; Odds Ratio (OR) = 1.31, 95% CI 2-sided [0.880 to 1.952]
Statistical Analysis 3: Comparison: Part A: Remdesivir for 5 Days vs Part A: SOC Therapy; Secondary analysis; Test type: Superiority; p = 0.0168, Proportional odds model — P-value was calculated using proportional odds model with treatment as the independent variable and baseline clinical status as a nominal covariate; Odds Ratio (OR) = 1.65, 95% CI 2-sided [1.095 to 2.497]
Statistical Analysis 4: Comparison: Part A: Remdesivir for 10 Days vs Part A: SOC Therapy; Secondary analysis; Test type: Superiority; p = 0.2186, Proportional odds model — [p-value comment as in outcome 1, analysis 3]; Odds Ratio (OR) = 1.29, 95% CI 2-sided [0.862 to 1.917]

2. Secondary Outcome: Part A: Percentage of Participants Who Experienced Treatment-Emergent Adverse Events (TEAEs)
Description: TEAEs were defined as the following: any AE with an onset date on or after the study treatment start date and no later than 30 days after permanent discontinuation of study treatment and/or any AE leading to premature discontinuation of study treatment. For participants randomized to the SOC group, all AEs reported on or after the protocol-specified Day 1 visit were considered as treatment emergent.
Time Frame: First dose date up to last dose date (maximum: 10 days) plus 30 days
Population: Safety Analysis Set included participants who were randomized into part A of the study and received at least 1 dose of study treatment or completed the Day 1 visit (SOC only group).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part A: Remdesivir for 5 Days | Part A: Remdesivir for 10 Days | Part A: SOC Therapy
Number analyzed (Participants) | 191 | 193 | 200
percentage of participants | 51.3 [44.0 to 58.6] | 58.5 [51.3 to 65.6] | 46.5 [39.4 to 53.7]
Statistical Analysis 1: Comparison: Part A: Remdesivir for 5 Days vs Part A: SOC Therapy; Test type: Superiority; p = 0.3633, Fisher Exact — P-value was calculated from the Fisher exact test to compare each RDV group and the SOC group; Difference in the Percentages = 4.8, 95% CI 2-sided [-5.2 to 14.7]
Statistical Analysis 2: Comparison: Part A: Remdesivir for 10 Days vs Part A: SOC Therapy; Test type: Superiority; p = 0.0201, Fisher Exact — P-value was calculated from the Fisher exact test to compare each RDV group and the SOC group; Difference in the Percentages = 12.0, 95% CI 2-sided [1.6 to 21.8]

ADVERSE EVENTS:
Time Frame: First dose date up to the last dose date (maximum: 10 days for Part A, 11 days for Part B) plus 30 days.
Description: Part A=Safety Analysis Set included participants who were randomized into part A of the study and received at least 1 dose of study treatment or completed the Day 1 visit (SOC only group); Part B=Expanded RDV-Treated Analysis Set included participants who were enrolled into part B of the study and received at least 1 dose of study drug.
Arm/Group | Part A: Remdesivir for 5 Days | Part A: Remdesivir for 10 Days | Part A: SOC Therapy | Part B: Extension Treatment, Remdesivir for 10 Days
All-Cause Mortality (participants affected / at risk) | 2/191 | 3/193 | 4/200 | 13/503
Serious Adverse Events (participants affected / at risk) | 9/191 | 10/193 | 18/200 | 40/503
Other Adverse Events (participants affected / at risk) | 41/191 | 42/193 | 30/200 | 113/503
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Remdesivir for 5 Days (N=191) | Part A: Remdesivir for 10 Days (N=193) | Part A: SOC Therapy (N=200) | Part B: Extension Treatment, Remdesivir for 10 Days (N=503)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 2 | 0
Cardiac failure acute (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 1
Death (General disorders) | 0 | 0 | 0 | 2
General physical health deterioration (General disorders) | 0 | 0 | 0 | 1
Impaired healing (General disorders) | 1 | 0 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 0 | 2
Pyrexia (General disorders) | 0 | 0 | 0 | 1
Arthritis infective (Infections and infestations) | 0 | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0
Biliary sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1
Corona virus infection (Infections and infestations) | 0 | 0 | 1 | 2
Empyema (Infections and infestations) | 0 | 0 | 0 | 1
Neutropenic sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 1
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia viral (Infections and infestations) | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Septic shock (Infections and infestations) | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 2
Post procedural bile leak (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0
Heart rate decreased (Investigations) | 1 | 0 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 2
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Brain oedema (Nervous system disorders) | 0 | 0 | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 1 | 0 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 1
Renal colic (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 2
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 5 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Lung opacity (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
Haemodynamic instability (Vascular disorders) | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 2
Shock (Vascular disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Remdesivir for 5 Days (N=191) | Part A: Remdesivir for 10 Days (N=193) | Part A: SOC Therapy (N=200) | Part B: Extension Treatment, Remdesivir for 10 Days (N=503)
Constipation (Gastrointestinal disorders) | 8 | 5 | 9 | 26
Diarrhoea (Gastrointestinal disorders) | 12 | 10 | 14 | 28
Nausea (Gastrointestinal disorders) | 19 | 18 | 6 | 41
Hypokalaemia (Metabolism and nutrition disorders) | 10 | 13 | 4 | 23
Headache (Nervous system disorders) | 10 | 10 | 5 | 27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (3):
  • Study Protocol (2020-04-29): https://cdn.clinicaltrials.gov/large-docs/30/NCT04292730/Prot_000.pdf
  • Statistical Analysis Plan: GS-US-540-5774-appendix-16.1.9-SAP part A_f-redact (2020-06-26): https://cdn.clinicaltrials.gov/large-docs/30/NCT04292730/SAP_001.pdf
  • Statistical Analysis Plan: GS-US-540-5774-appendix-16.1.9-SAP part B_f-redact (2020-09-16): https://cdn.clinicaltrials.gov/large-docs/30/NCT04292730/SAP_002.pdf